CLINICAL TRIAL: NCT05041387
Title: Data Collection of Standard Care of Patients in the EMG Section
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000560; 000560-N
Record Dates: First submitted 2021-09-10; First posted 2021-09-13 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09-12

CONDITIONS: Neuropathy; Muscle Disorders; Dysautonomia
Keywords: Standard of Care; Screening; NEUROMUSCULAR DISORDERS
MeSH Terms: conditions — Muscular Diseases; Autonomic Nervous System Diseases; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neuromuscular disorders: Patients with neuromuscular disorders, no specific diagnosis

SUMMARY:
Background:

Most people who are referred to the EMG (Electromyography) Section of the NIH are enrolled into specific active studies. This allows researchers to learn about a range of rare neuromuscular disorders. But study criteria may not give researchers the chance to evaluate a single person or study a common symptom. Therefore, researchers want to assess people with neuromuscular disorders who are not currently enrolled in any NIH studies. They will perform tests on these individuals in the EMG Lab. Then they will create a repository of data that may be used for future research. This will help them learn more about these disorders.

Objective:

To retain data that is collected as part of participant visits to the NIH.

Eligibility:

People aged 18 and older who will be visiting the NIH for evaluation of their neuromuscular disorder.

Design:

Participants will be screened with a medical record review.

Participants will have a physical exam. They will be evaluated for their neuromuscular disorder. They may have tests to learn more about how their nerves and muscles work that are called nerve conduction and EMG studies. Their muscles and nerves may be assessed with an ultrasound. Their ability to sweat may be measured. Their heart rate and blood pressure may be taken. Changes to their breathing or changes in their body position may be measured.

Participant data will be given a unique numerical identifier that can be used if the data is shared. Data will be stored on a server and in a database.

Participants will have 1-2 visits. Each visit will last less than 4 hours. They may be contacted for a follow-up visit.

DETAILED DESCRIPTION:
Study Description:

This protocol is designed to create a repository of information for future hypothesis generation. We will be evaluating patients with neuromuscular disorders that are not currently enrolled in any NIH protocols with procedures performed in the EMG Lab. The procedures include standard neurophysiological studies of EMG, autonomic nervous system (ANS) testing, and neuromuscular ultrasound (NMUS) as deemed necessary for appropriate diagnostic and clinical status testing. This will allow us to investigate into the problems of these patients with the purpose of furthering general knowledge of neuromuscular disorders and enhancing our EMG capabilities. Our ability to evaluate patients with a wide variety of neuromuscular diseases is also critical to maintaining our accreditation with the clinical neurophysiology fellowship programs and training our fellows to be competent physicians, as well as for keeping all staff, including senior staff, up-to-date and familiar with the evaluation of patients with a wide spectrum of diseases. We may also be able to later refer these patients into treatment protocols or re-evaluate patients that are no longer in an active NINDS protocol. This protocol will be valuable resource to the community by engendering greater interaction with the local neurologists and clinics as well as providing certain types of neurophysiological testing that are not readily available in the community.

Objectives:

To create a repository of information on enrolled participants to allow for hypothesis generation in future research

To add value to the Clinical Neurophysiology training programs by providing consult, diagnostic tests, and medical follow-up of participants

Endpoints:

To create a repository of information on enrolled participants to allow for hypothesis generation in future research.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* The patient or the patient's Legally Authorized Representative is capable of informed consent and signs the consent form.
* Male or female, age 18 and over, no age limit
* Possible neuromuscular disorder or neurodegenerative disorder.

EXCLUSION CRITERIA:

No other exclusion criteria for patients

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be referred by physician, clinic or may be self-referred.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2031-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
To provide a repository of information on enrolled participants to allow for hypothesis generation in future research. | 10 years
  Results of patient's studies will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya J Lehky, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be shared with the referring physician and any other person the participant requests. The individual participant data will not be shared with anyone not involved in the care of that participant.
Supporting Information: CSR
Time Frame: As mentioned above, IPD will only be shared with the referring physician.
Access Criteria: No analysis or general data will be shared.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000560-N.html